CLINICAL TRIAL: NCT02062606
Title: Preservation of Thoracic Kyphosis and Coronal Curve Correction as a Function of Rod Stiffness in the Surgical Treatment of Adolescent Idiopathic Scoliosis (AIS) With the Use of the K2M MESA Rail™ Deformity System
Brief Title: MESA Rail™ AIS Study - Preservation of Curve Correction
Status: Terminated | Type: Observational
Why Stopped: The study terminated early due to slow enrollment that significantly extended the expected study duration.
Sponsor: K2M, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-001
Record Dates: First submitted 2014-01-31; First posted 2014-02-13 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Spinal Curvatures; Spinal Diseases; Adolescent Idiopathic Scoliosis; Spinal Deformity
MeSH Terms: conditions — Scoliosis; Spinal Curvatures; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AIS: Surgical implantation of the K2M MESA Rail™ Deformity System in the treatment of Adolescent Idiopathic Scoliosis (AIS).
  Interventions: Device: MESA Rail™ Deformity System

INTERVENTIONS:
Device: MESA Rail™ Deformity System — MESA Rail™ (cross-sectioned rod) with MESA pedicle screws compared to traditional rod use in the literature

SUMMARY:
To evaluate the restoration and maintenance of thoracic kyphosis and coronal curve correction demonstrated through the surgical implantation of the K2M MESA Rail™ Deformity System as compared to literature reported outcomes for standard Cobalt Chrome (CoCr) rod systems in the treatment of Adolescent Idiopathic Scoliosis (AIS).

DETAILED DESCRIPTION:
Patients treated with the Ø5.5mm or Ø4.5mm MESA Rail™ Deformity System that had:

Diagnosis of AIS requiring surgical treatment for selective non-cervical fusion with a minimum of five (5) instrumented vertebrae between T1-S1 as confirmed by patient history and radiographic studies.

AIS cases must be classified as a Lenke type 1 or type 2 curve (lumbar modifiers and thoracic sagittal profiles will be noted but not restrictive).

Age at time of surgery of ≥ 11 years old and ≤ 21 years old.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS requiring surgical treatment for selective thoracic/lumbar fusion with a minimum of five (5) instrumented vertebrae between T1-S1 as confirmed by patient history and radiographic studies. AIS cases must be classified as a Lenke type 1 or type 2 curve. No cervical vertebrae are to be incorporated into the construct.
* Willingness and ability to comply with the requirements of the protocol including follow-up requirements.
* Willing and able to sign a study specific informed consent form or, in the case of a patient who is a minor, provide assent and the minor patient's parent/legal guardian provides written consent to participate.
* Age range of ≥ 11 years old and ≤ 21 years old at time of surgery.

Exclusion Criteria:

* Previous anterior or posterior spine surgery at the index levels.
* Previous posterior spine surgery (e.g., posterior element decompression) that destabilizes the cervical/thoracic/lumbar spine.
* Active systemic infection or infection at the operative site.
* Co-morbid medical conditions of the spine or upper/lower extremities that may affect the thoracic or lumbar spine neurological and/or pain assessment.
* Metabolic bone disease such as osteoporosis that contradicts spinal surgery.
* History of an osteoporotic fracture.
* History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism.
* Taking medications that may interfere with bony/soft tissue healing including chronic steroid use.
* Known allergy to titanium or cobalt chrome.
* Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia.
* Insulin-dependent type 1 or type 2 diabetes.
* Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion.
* Pregnant, or intend to become pregnant, during the course of the study.
* Severe obesity (Body Mass Index > 40).

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Two-hundred four (204) total subjects with the MESA Rail Deformity System at up to 18 clinical sites, geographically distributed worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2014-05; Primary Completion 2020-02-23 (Actual); Study Completion 2020-02-23 (Actual)

REFERENCES:
- [Background] Wattenbarger JM, Richards BS, Herring JA. A comparison of single-rod instrumentation with double-rod instrumentation in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2000 Jul 1;25(13):1680-8. doi: 10.1097/00007632-200007010-00011. PMID 10870143
- [Background] Newton PO, Yaszay B, Upasani VV, Pawelek JB, Bastrom TP, Lenke LG, Lowe T, Crawford A, Betz R, Lonner B; Harms Study Group. Preservation of thoracic kyphosis is critical to maintain lumbar lordosis in the surgical treatment of adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2010 Jun 15;35(14):1365-70. doi: 10.1097/BRS.0b013e3181dccd63. PMID 20505560
- [Background] Kim YJ, Lenke LG, Bridwell KH, Kim J, Cho SK, Cheh G, Yoon J. Proximal junctional kyphosis in adolescent idiopathic scoliosis after 3 different types of posterior segmental spinal instrumentation and fusions: incidence and risk factor analysis of 410 cases. Spine (Phila Pa 1976). 2007 Nov 15;32(24):2731-8. doi: 10.1097/BRS.0b013e31815a7ead. PMID 18007253

RESULTS

PARTICIPANT FLOW:
Groups:
- K2M MESA Rail™ Deformity System: Patients treated with the Ø5.5mm or Ø4.5mm MESA Rail Deformity System that had:
  1. Diagnosis of AIS requiring surgical treatment for selective thoracic/lumbar fusion with a minimum of five (5) instrumented vertebrae between T1-S1 as confirmed by patient history and radiographic studies. AIS cases must be classified as a Lenke type 1 or type 2 curve (lumbar modifiers and thoracic sagittal profiles were noted but not restrictive).
  2. An age at time of surgery of ≥ 11 years old and ≤ 21 years old
Period: Overall Study
Arm/Group | K2M MESA Rail™ Deformity System
Started | 188
Completed | 99
Not Completed | 89

BASELINE CHARACTERISTICS:
Groups:
- Demographics and Baseline Characteristics: This is a demographic and baseline characteristics of the patient population. This includes parameters such as Age, Gender, Height, Weight Body Mass Index (BMI) and Tobacco Usage.
Arm/Group | Demographics and Baseline Characteristics
Number analyzed (Participants) | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 180
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.65 (2.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study Case Report Forms did not include Race/Ethnicity
Region of Enrollment [Number; unit: participants]
  United States | 170
  New Zealand | 4
  Australia | 14
Height [Mean (Standard Deviation); unit: cm] | 160.4 (10.8)
Weight [Mean (Standard Deviation); unit: kg] | 55.3 (13.53)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.43 (4.66)
Tobacco Use [Count of Participants; unit: Participants]
  Never | 186
  Quit | 1
  Currently Use | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Thoracic Kyphosis and Coronal Curve Correction on X-ray at 24 Months
Description: Restoration and maintenance of thoracic kyphosis and coronal curve correction.
  Thoracic kyphosis (Coronal Curve): measurement of curvature from the upper endplate of T4 to the lower endplate of T12.
Time Frame: Baseline (up to 90 days before surgery), 24 months
Population: 98 of the 99 participants who returned at 24 Months had the thoracic kyphosis measurement.
Measure: Mean (95% Confidence Interval); unit: degrees
Groups:
- All Patients: The overall change of Thoracic Kyphosis (TK) within the current study.
Arm/Group | All Patients
Number analyzed (Participants) | 98
degrees | -3.84 [-5.91 to -1.76]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with SAE and AE for the various intervals
Time Frame: Up to 24 months
Population: This is an analysis of the number of participants that reported any form of adverse event. Overall participants with any AE or SAE. 5 of the 17 SAE participants did not experience a non-SAE events. The other 12 participants had events in both categories. The study did not establish a frequency threshold, therefore, all AEs are listed.
Measure: Number; unit: participants
Groups:
- Up to Post-Operative; Post-Operative to 3 Months; 3 to 6 Months; 6 to 12 Months; 12 to 24+ Months: participants with SAE and AE
- Overall: Overall number of participants with SAE and AEs
Arm/Group | Up to Post-Operative | Post-Operative to 3 Months | 3 to 6 Months | 6 to 12 Months | 12 to 24+ Months | Overall
Number analyzed (Participants) | 188 | 160 | 147 | 135 | 99 | 188
participants
  Any AE | 62 | 7 | 21 | 25 | 36 | 98
  Any AE : Procedure Related | 44 | 0 | 12 | 9 | 18 | 67
  Any AE : Device Related | 16 | 0 | 3 | 6 | 7 | 26
  Any AE : Mild | 44 | 6 | 17 | 20 | 29 | 79
  Any AE : Moderate | 19 | 1 | 4 | 5 | 10 | 31
  Any AE : Severe | 5 | 1 | 0 | 1 | 0 | 7
  Any SAE | 10 | 1 | 0 | 4 | 3 | 17
  Any SAE : Procedure Related | 8 | 0 | 0 | 1 | 2 | 11
  Any SAE : Device Related | 2 | 0 | 0 | 1 | 2 | 5
  Any SAE : Mild | 3 | 0 | 0 | 1 | 1 | 5
  Any SAE : Moderate | 4 | 0 | 0 | 2 | 2 | 7
  Any SAE : Severe | 4 | 1 | 0 | 1 | 0 | 6

3. Secondary Outcome: Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at 24 Months
Description: Evaluation of the improvement of the Back VAS and Hip/Leg VAS (assessed together) at the 24 month post-operative visit as compared to pre-op time periods. Information on all reports of pain/numbness /tingling and the location of symptoms were captured and evaluated.
  VAS scale ranged from 0 - 100mm with the 100mm accounting for the highest level of pain.
Time Frame: Baseline (up to 90 days before surgery), 24 months
Population: 13 out of the 99 participants who returned at 24 months, did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Back; Left Leg/Hip; Right Leg/Hip: pain scores on the VAS
Arm/Group | Back | Left Leg/Hip | Right Leg/Hip
Number analyzed (Participants) | 86 | 86 | 86
score on a scale | -16.9 (29.5) | -0.2 (13.2) | -2 (17.8)

4. Secondary Outcome: Change From Baseline in Quality of Life Scores on the SRS-22r at 24 Months
Description: The Revised Scoliosis Research Society-22 (SRS-22r) is a specific questionnaire for spine conditions. It is applied to patients with idiopathic scoliosis, whose conditions and treatments have a great impact on their quality of life. The SRS 22r was created and revised with the purpose of evaluating this impact from the patient's point of view. The reviewed version contains 22 questions distributed into five domains: function/activity (FA), pain (P), self- image/appearance (SA), mental health (MH) and satisfaction with treatment (ST).
  The scores vary from 1 to 5 in which 5 is the best health quality of life of patients.
Time Frame: Baseline (up to 90 days before surgery), 24 months
Population: While 99 participants completed 24 month interval, 14 patients out of the 99 did not did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 24 Month: Baseline in quality of life scores on the SRS-22r
Arm/Group | 24 Month
Number analyzed (Participants) | 85
score on a scale | 0.6 (0.7)

5. Secondary Outcome: Patient Satisfaction
Description: At the 12 month and 24 month follow-up visits, subjects were asked whether they were satisfied with the outcome of their surgery (Yes/No) and whether they would repeat the operation (Yes/No).
Time Frame: 12 months and 24 months
Population: Patient self-assessment of the procedure at 12M and 24M
Measure: Count of Participants; unit: Participants
Groups:
- 12 Month; 24 Month: Patient satisfaction at 12 Month
Arm/Group | 12 Month | 24 Month
Number analyzed (Participants) | 135 | 99
Participants
  Satisfied: Yes | 124 | 86
  Satisfied: No | 4 | 2
  Satisfied: Not Reported | 7 | 11
  Repeat Procedure: Yes | 105 | 76
  Repeat Procedure: No | 23 | 12
  Repeat Procedure: Not Reported | 7 | 11

6. Secondary Outcome: Investigator's Rating of Subject's Clinical Disposition Using Odom's Criteria
Description: At the 24 month follow-up visit, the Investigator rated the clinical disposition of each study subject according to Odom's Criteria as follows:
  Excellent: all pre-operative symptoms relieved, able to carry out daily occupations without impairment.
  Good: minimum persistence of pre-operative symptoms, able to carry out daily occupations without significant interference.
  Fair/Satisfactory: relief of some pre-operative symptoms but physical activity is significantly limited.
  Poor: symptoms or signs unchanged or worsened.
Time Frame: 24 months
Population: Patients who were rated based on the outcome of their treatment and would indicate either Excellent, Good or Fair/Satisfactory. No responses are shown under missing
Measure: Count of Participants; unit: Participants
Groups:
- Investigator's Rating: Investigator's rating of subject's clinical disposition using Odom's Criteria
Arm/Group | Investigator's Rating
Number analyzed (Participants) | 99
Participants
  Fair/Satisfactory | 2
  Good | 15
  Excellent | 78
  Missing | 4

7. Secondary Outcome: Length of Surgery Time
Description: The length of the surgical procedure from the initial incision to final closure were captured.
Time Frame: During surgery
Population: 186 patients had their surgery times recorded. There were 3 additional procedures staged increasing the overall number of units analyzed to 189.
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: surgeries
Groups:
- Length of Surgery Time: The length of the surgical procedure from the initial incision to final closure
Arm/Group | Length of Surgery Time
Number analyzed (Participants) | 186
Number analyzed (surgeries) | 189
Minutes | 267.01 (79.89)

8. Secondary Outcome: Length of Anesthesia Time
Description: The length of time the patient is under anesthesia was captured.
Time Frame: During surgery
Population: 183 subjects had anesthesia time included. There were 3 staged procedures increasing the overall number of units analyzed to 186.
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: surgeries
Groups:
- Length of Anesthesia Time: The length of time the patient is under anesthesia was captured.
Arm/Group | Length of Anesthesia Time
Number analyzed (Participants) | 183
Number analyzed (surgeries) | 186
Minutes | 373.67 (91.97)

9. Secondary Outcome: Estimated Blood Loss
Description: The amount of blood loss over the entire length of the surgery was captured.
Time Frame: During surgery
Population: 187 patients had blood loss included. There were 3 additional procedures staged increasing the overall number of units analyzed to 190.
Measure: Mean (Standard Deviation); unit: Cubic Centimeters
Units Other Than Participants: surgeries
Groups:
- Estimated Blood Loss: The amount of blood loss over the entire length of the surgery was captured.
Arm/Group | Estimated Blood Loss
Number analyzed (Participants) | 187
Number analyzed (surgeries) | 190
Cubic Centimeters | 672.34 (588.14)

10. Secondary Outcome: Length of Hospital Stay
Description: The length of the hospital stay from the date of admission to the date of discharge.
Time Frame: Admission to Discharge
Population: 186 patients completed admit and discharge dates
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: surgeries
Groups:
- Length of Hospital Stay: The length of the hospital stay from the date of admission to the date of discharge
Arm/Group | Length of Hospital Stay
Number analyzed (Participants) | 186
Number analyzed (surgeries) | 186
Days | 5.28 (1.79)

11. Secondary Outcome: Change in Percentage of Participants Able to Return to Work/School
Description: The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery by looking at the change in percentage of participants who were able to return to work without any restrictions
Time Frame: Pre-Op to 24 months
Population: Includes all participants who returned for each visit interval with those who did not respond to this question accounted for in the missing row.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Op; Initial Post Op; 3 Month; 6 Month; 12 Month; 24 Month: The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery was documented.
Arm/Group | Pre-Op | Initial Post Op | 3 Month | 6 Month | 12 Month | 24 Month
Number analyzed (Participants) | 188 | 181 | 160 | 147 | 135 | 99
Participants
  Unemployed, unrelated to back/leg conditions | 0 | 0 | 0 | 0 | 0 | 0
  Not attending work/school by choice | 11 | 22 | 7 | 2 | 3 | 0
  Unable to go due to back/leg pain/conditions | 0 | 57 | 4 | 0 | 0 | 0
  Attending work/school with some restrictions | 5 | 83 | 104 | 44 | 14 | 4
  Attending work/school with no restrictions | 172 | 19 | 44 | 101 | 117 | 93
  Missing | 0 | 0 | 1 | 0 | 1 | 2

12. Secondary Outcome: Use of Narcotics Post-surgery
Description: The types and dosages of any narcotics taken by the patient pre- and post-surgery was documented.
Time Frame: Pre-Op to 24 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Op; Initial Post Op; 3 Month; 6 Month; 12 Month; 24 Month: The types and dosages of any narcotics taken by the patient pre- and post-surgery was be documented.
Arm/Group | Pre-Op | Initial Post Op | 3 Month | 6 Month | 12 Month | 24 Month
Number analyzed (Participants) | 188 | 181 | 160 | 147 | 135 | 99
Participants
  Back Meds: None | 128 | 46 | 118 | 114 | 112 | 78
  Back Meds: Non-narcotics or NSAIDS | 53 | 28 | 29 | 28 | 22 | 16
  Back Meds: Intermittent short-acting narcotics | 6 | 77 | 9 | 5 | 1 | 1
  Back Meds: Chronic daily short-acting narcotics | 1 | 18 | 2 | 0 | 0 | 0
  Back Meds: Chronic daily long-acting narcotics | 0 | 6 | 1 | 0 | 0 | 0
  Back Meds: IV or injected narcotics | 0 | 6 | 0 | 0 | 0 | 0
  Back Meds: Epidural/Facet injection | 0 | 0 | 0 | 0 | 0 | 0
  Back Meds: Missing | 0 | 0 | 1 | 0 | 0 | 4
  Non-Back Meds: None | 157 | 151 | 141 | 125 | 118 | 84
  Non-Back Meds: Non-narcotics or NSAIDS | 31 | 22 | 18 | 22 | 17 | 13
  Non-Back Meds: Intermittent short-acting narcotics | 0 | 7 | 0 | 0 | 0 | 0
  Non-Back Meds: Chronic daily short-acting narcotics | 0 | 1 | 0 | 0 | 0 | 0
  Non-Back Meds: Chronic daily long-acting narcotics | 0 | 0 | 0 | 0 | 0 | 0
  Non-Back Meds: IV or injected narcotics | 0 | 0 | 0 | 0 | 0 | 0
  Non-Back Meds: Epidural/Facet injection | 0 | 0 | 0 | 0 | 0 | 0
  Non-Back Meds: Missing | 0 | 0 | 1 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: From Operative to 24+ Months
Description: Any untoward medical occurrence in a subject undergoing surgery in this trial which does not necessarily have a causal relationship with this intervention. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the one of the devices. Any AE that occurs during the subject's participation in the study will be recorded on the Adverse Event case report form.
Groups:
- Participants With Adverse Events: Overall participants with any AE or SAE.
  5 of the 17 SAE participants did not experience a non-SAE events. The other 12 participants had events in both categories.
  The study did not establish a frequency threshold, therefore, all AEs are listed.
Arm/Group | Participants With Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/188
Serious Adverse Events (participants affected / at risk) | 17/188
Other Adverse Events (participants affected / at risk) | 93/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=188)
Infectious mononucleosis (Blood and lymphatic system disorders) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Complications associated with device (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 3 (3)
Sensory loss (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=188)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Infectious mononucleosis (Blood and lymphatic system disorders) | 1 (2)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Salivary gland mucocoele (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Chest pain (General disorders) | 10 (11)
Chills (General disorders) | 1 (1)
Complication associated with device (General disorders) | 4 (5)
Cyst (General disorders) | 2 (2)
Flank pain (General disorders) | 2 (2)
Hypertrophy (General disorders) | 1 (1)
Pain (General disorders) | 16 (20)
Pyrexia (General disorders) | 4 (4)
Respiratory complication associated with device (General disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (2)
Viral pharyngitis (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 7 (12)
Incision site discharge (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Body temperature decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (30)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal apin (Musculoskeletal and connective tissue disorders) | 15 (18)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysaesthesia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 8 (9)
Migraine (Musculoskeletal and connective tissue disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 3 (4)
Neuralgia (Nervous system disorders) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (3)
Poor quality sleep (Nervous system disorders) | 1 (1)
Spinal muscular atrophy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Vertigo (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Body tinea (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Kerion (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution/PI shall not disclose/use any confidential/proprietary information (CI) disclosed to/developed by the Institution during the study. Institution/PI agree to hold the results of the Study in confidence, and shall not disclose them except with prior written consent of K2M. Institution agrees to submit any Articles to K2M for review prior to publication and agrees to edit out any confidential information identified by K2M.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT02062606/Prot_SAP_000.pdf